CLINICAL TRIAL: NCT00175201
Title: From Efficacy to Effectiveness of a Proactive Perioperative Care and Rehabilitation in Patients Undergoing Primary Total Hip or Knee Replacement
Brief Title: Cost Efficacy of a Clinical Pathway to Patients Undergoing Hip and Knee Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KL-05-01
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Rehabilitation

INTERVENTIONS:
Procedure: Proactive care and rehabilitation

SUMMARY:
In this randomised study a proactive care and rehabilitation intervention is compared to the current care and rehabilitation in patients undergoing primary hip and knee replacement surgery.

A cost efficacy analysis in a societal perspective is made from effect data in the randomised controlled study together with cost data gathered during the perioperative and postoperative period.

If the proactive care and rehabilitation intervention is cost effective the intervention is going to be implemented in Ringkøbing County. This implementation proces is measured within a monitoring project of all patients receiving hip or knee replacement surgery in Ringkøbing County in the period 2003 to 2007.

DETAILED DESCRIPTION:
BACKBROUND Hip and knee replacement are commonly performed surgical procedures, with more than 800,000 hip operations carried out worldwide each year and with almost 550 hip and knee replacements each year in Ringkoebing County. The main indicators for total hip or knee replacement are intractable pain and/or limitation of function that cannot be managed by conservative treatment alone. Leading causes of such pain include osteoarthritis, rheumatoid arthritis, trauma, congenital abnormalities, dysplasia and osteochondritic disease. In the absence of treatments that provide a cure for conditions such as osteoarthritis, management is directed primarily towards relieving pain and re-ducing functional limitation. Joint replacement is one surgical option when medical treatment has failed to provide adequate symptom relief. Hip or knee replacement is a major surgical procedure that requires inpatient physiotherapy and out-patient rehabilitation following a stay in hospital.

Regarding the effect of optimizing the perioperative period, no systemically critical reviews of randomized controlled trials (RCT) could be identified. Only one RCT of the effect of a clinical pathway in hip and knee arthroplasty could be identified, the study by Dowsey et al from 1999, which concludes that the intervention gives a better effect and reduces the average length of stay with 1.5 day. No cost data were reported in this study. A systematic review of clinical pathways including the study by Dowsey et al and ten non-RCT studies concludes that clinical pathways for total knee and total hip arthroplasty reduces costs and length of stay. A significant and great reduction in length of stay is reported from two resent Danish non-RCT, the study by Rasmussen et al, in which an accelerated and proactive care was given and the study by Husted et al, in which no extra resources were allocated but the care was given in a special unit focusing on a length of stay of maximal 8 days. However nothing is known about the cost or effects of this accelerated and proactive care out-side the hospital.

In summary the overall evidence level on accelerated perioperative care and rehabilitation for patients undergoing total hip or knee replacement is scarce.

OBJECTIVES To investigate the cost efficacy of a focused and specialized care unit in patients undergoing total hip or knee replacement

To investigate the cost effectiveness of a focused and specialized care unit in patients under-going total hip or knee replacement

MATERIALS & METHODS: Randomized controlled intervention trial with cost efficacy and cost effectiveness analysis. This study follows the recommendations by the CONSORT Statement.

Perioperative study - RCT Study subjects All patients planned to undergo a primary total hip or total knee replacement at the Hospital in Holstebro, are at first contact to the hospital invited to participate in the study. Exclusion criteria's are patients operated secondary to a hip fracture, patients undergoing remission and patients who are not able to cooperate normally during the perioperative period. All patients interested in participating in the study are given written and oral information. After consent the participating patients completes a baseline questionnaire and are randomized to one of the two groups.

Sample size The estimated sample size of the groups at followup was calculated using actual data from the hospital in Holstebro from the year 2004 together with data from a pilot study in 2005. The risk of performing a Type 1 error was set at 5% using a two-sided analysis, and the power of detecting a true difference was set at 80%. The anticipated reduction of length of stay was set at 2 days in the intervention group, from a mean length of stay of 8 days with a standard deviation (SD) of 4 days to a mean length of stay of 6 days and SD of 2 days. When using a two-sample comparison of means this gives a need for at least 80 patients, 40 persons in each group at follow-up.

Randomization Simple randomization ensuring equal distribution of operation area (hip:knee) is performed by drawing an envelope from a box.

Intervention Control group Patients in the control group receive the current perioperative care.

Intervention group Patients in the intervention group are given perioperative care and rehabilitation according to the regime advocated by The Unit for Perioperative Nursing Care,Rigshospitalet and in the study by Husted et al and. In this study the perioperative care and rehabilitation is organized in a new proactive special care and rehabilitation unit where the patients are gathered and the health care staff are focusing on a preselected discharge day.

Attempts to reduce potential bias Masking of the patients is obtained by concealment of the intervention in the other intervention groups, and by securing that the patients in the two different groups are kept apart in different rooms. Masking of the treating therapists and caretaking nurses are attempted by randomly allocating them to either usual or the new preoperative care and rehabilitation unit. All personal allocated to the new preoperative unit receive education and participates in a pre study period. After starting the intervention period the treating therapists and caretaking nurses are not allowed to attend the rooms of patients not allocated to their intervention arm. During the intervention period physiotherapists and nurses are not allowed to discuss the intervention with persons in the other intervention arm. Situation and circumstances where the protocol is not followed will be registered using an intervention log book. The baseline and follow-up data collection is performed with questionnaires and by measurements by a person not involved in the intervention. No attempt is made to minimize the placebo or the Hawthorne effect, because the different attention and time spent in the intervention is an important factor in the cost effectiveness analysis. Potential contamination regarding the care given by nurses and treating therapists is recorded via a structured observation of care and treatment before baseline and in the latter part the study period. Compliance with exercise is collected through the reporting of actual participation in planned training and questionnaires filled inat day of discharge.

Follow-up Length of stay is recorded using register information and all other outcome measures are collected from questionnaires at discharge, 3, 12 and 24 months after discharge.

Outcome measures Primary outcome measures are length of stay, health related quality of life measured with EQ-5D and SF-36/SF-6D. Secondary outcome measures are pain measured with a 6/point ordinal scale, disability measured with Harris Hip Score / The Danish Knee Arthroplasty Register Score.

Side effects are collected from register data on mortality and the incidence and length of stay be-cause of deep vein thrombosis.

Data analysis The data is analysed according to the recommendations by Sackett et al using intention-to-treat analysis. Chi-square test is used for categorical data and parametric or non-parametric statistics for two-sample comparison of means are used for continuous data. The significance level is set at p<0.05.

Cost efficacy study of a perioperative intervention Efficacy is in this study defined according to Last JM as: The extent to which a specific intervention, procedure, regimen, or service produces a beneficial result under ideal conditions. Ideally, the determination of efficacy is based on the results of a randomized controlled trial. The question to be answered according to Drummond MF et al is: Can it work? To determine whether a proactive perioperative intervention in patients undergoing total hip or knee replacement is cost effective under ideal circumstances the study is performed alongside the RCT at one hospital. Actual costs are sought via available data sources and patient administered diaries and collected for a period of 24 months. The collected cost data are divided into direct costs and benefits, indirect costs and benefits and intangible costs and benefits. Direct healthcare costs include peripoperative operation and hospital stay costs at DRG taxes together with changes in costs due to the perioperative intervention at actual prices. Direct postoperative primary health care sector costs include costs from visiting general practitioner, nurses and physiotherapist at preset prices. Direct non-healthcare costs includes social sector costs such as professional home care and extra costs at nursery homes, private home care costs, private rehabilitation costs, costs from visiting alternative therapists, private help costs and transportation costs at preset prices. Indirect costs are costs from production loss and are estimated according to the friction method with a maximum of 3 months of absenteeism from paid work at preset salary. Intangible costs and benefits are not collected beneath being implicit in the quality of life measures. The costs are held against the primary outcome measures in each group. The cost efficacy of the intervention is calculated as the differences in costs related to the differences in effects between the intervention and control group. The cost efficacy analysis is performed according to the recommendations by Drummond et al.

Cost effectiveness study of a perioperative intervention Effectiveness is in this study defined according to Last JM as: The extent to which a specific intervention, procedure, regimen, or service, when deployed in the field of routine circumstances, does what it is intended to do for a specific population. The question to be answered according to Drum-mond MF et al is: Does it work? To determine whether a proactive perioperative intervention in patients undergoing total hip or knee replacement is cost effective in other units in the county under normal circumstances the estimated cost difference from the efficacy study together with the im-plementation time, problems and costs of the fully developed intervention is held against the actual effect difference of all outcome measures for the period following implementation compared the period prior to implementation. The cost effectiveness analysis is performed according to the recommendations by Drummond et al.

ELIGIBILITY:
Inclusion Criteria:

Primary osteoarthritis of the hip and knee -

Exclusion Criteria:

Non-cooperative Replacement secondary to fracture Revision surgery

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2006-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Health relatede quality of life
Pain
Disabillity
Costs

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, DMSC, Study Chair — Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Kristian Larsen, Holstebro, Jutland, Denmark